CLINICAL TRIAL: NCT07269847
Title: A Randomized Study to Compare the Effect of a Healthy Beef-Centric Diet to a Healthy U.S.-Style Dietary Pattern on Inflammation and Other Metabolic Health Outcomes in a Metabolic Syndrome and/or Pre-Diabetic Population
Brief Title: Comparing a Healthy Beef-Centric Diet to a Healthy U.S.-Style Diet on Metabolic Health Outcomes in Pre-Diabetic Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B06-25-01-T0086
Record Dates: First submitted 2025-11-14; First posted 2025-12-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Syndrome (MetS); Inflammation; Pre-Diabetes; Overweight or Obese Adults
Keywords: Healthy Beef-Centric Diet; Healthy U.S.-Style Dietary Pattern; Inflammation; Metabolic Syndrome; Pre-Diabetes
MeSH Terms: conditions — Metabolic Syndrome; Inflammation; Glucose Intolerance; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy U.S.-Style Dietary Pattern (Active Comparator): This diet is based on USDA's MyPlate dietary guidelines and includes a balanced intake of fruits, vegetables, whole grains, lean proteins, and low-fat dairy. This diet reflects a conventional, guideline-based approach to healthy eating.
  Interventions: Other: Healthy U.S.-Style Dietary Pattern
- Healthy Beef-Centric Diet (Experimental): This is a whole-food dietary pattern that emphasizes beef as the primary source of protein. This diet is designed to reflect a low-carbohydrate, minimally processed eating pattern.
  Interventions: Other: Healthy Beef-Centric Diet

INTERVENTIONS:
Other: Healthy Beef-Centric Diet — The TD is a whole-food dietary pattern that emphasizes beef as the primary source of protein. This diet is designed to reflect a low-carbohydrate, minimally processed eating pattern.
  Other Names: Test Diet (TD)
  Arms: Healthy Beef-Centric Diet
Other: Healthy U.S.-Style Dietary Pattern — The CD is based on the USDA's MyPlate dietary guidelines and includes a balanced intake of fruits, vegetables, whole grains, lean proteins, and low-fat dairy. The CD reflects a conventional, guideline-based approach to healthy eating.
  Other Names: Comparator Diet (CD)
  Arms: Healthy U.S.-Style Dietary Pattern

SUMMARY:
This randomized study will be conducted to compare the effect of a healthy beef-centric diet to a healthy U.S.-style dietary pattern on inflammation and other metabolic health outcomes in a metabolic syndrome and/or pre-diabetic population.

DETAILED DESCRIPTION:
This study follows a randomized, open-label, parallel design to compare the effects of a healthy beef-centric diet to a healthy U.S.-style dietary pattern on inflammation and other metabolic health outcomes in a metabolic syndrome and/or pre-diabetic population.

The comparator diet in this study is a U.S. Department of Agriculture (USDA) Healthy U.S.-Style Dietary Pattern, as outlined in the 2020 Dietary Guidelines for Americans, which emphasizes the consumption of nutrient-dense foods across all food groups in recommended amounts. This includes a variety of vegetables, fruits, whole grains, low-fat dairy, lean protein sources, and healthy oils, while limiting added sugars, saturated fats, and sodium.

The test diet in this study involves a healthy beef-centric diet, where beef is the main source of protein. Participants will consume 70% of their daily energy intake from beef. The rest of their calories will come from other protein and fat sources (20%), along with a small amount (10%) from low-carbohydrate fruits (such as berries) and vegetables (like dark leafy greens). This diet excludes all grains. While the carbohydrate intake is low, it is slightly higher than that of a typical ketogenic diet.

The healthy beef-centric diet is being investigated for its effects on metabolic health after a 5 week intervention period. This study will investigate whether a beef-centric diet will support management of glycemic control, inflammation, and lipid-related risk factors, while also enhancing quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 - 64 years of age (inclusive) at the time of signing the informed consent.
* Have a BMI range of 25.0 - 39.9 kg/m2 (inclusive).
* In otherwise generally good health as determined by the investigator.
* Have blood hs-CRP levels equal to or greater than 2.0 mg/L at screening.
* Have the following conditions at screening:

  1. Pre-diabetes (defined as an HbA1c of 5.7-6.4% [inclusive]), and/or
  2. MetS, i.e., have 3 of the 5 following metabolic criteria:

     * A waist circumference of more than 40 inches (102 cm) in men and 35 inches (88 cm) in women
     * Serum triglycerides level of 150 mg/dL (1.7 mmol/L) or greater
     * Reduced HDL cholesterol, less than 40 mg/dL (1.0 mmol/L) in men or less than 50 mg/dL (1.3 mmol/L) in women
     * Elevated fasting glucose of 100 mg/dL (5.6 mmol/L) or greater
     * Blood pressure values of systolic 130 mmHg or higher or diastolic 85 mmHg or higher
* Report low levels of physical activity, as defined by a "low" activity classification on the IPAQ-SF.
* Consume meat-based protein as a part of their normal diet and regularly consume beef.
* Not currently using, defined as ≤ 3 uses in the past 3 months prior to Visit 2, any nicotine containing products (patches, gums, vapes, etc.), and willing to abstain for 14 days before Visit 2 until the last procedure.
* Have maintained a stable, self-reported body weight for at least 6 months prior to screening (maximum ±10% change in self-reported body weight).
* Willing and able to consume all aspects of either study dietary intervention.
* Willing to adhere to all study dietary intervention prohibitions and restrictions.
* Have maintained consistent dietary habits, including medication and supplement intake, and lifestyle for the last 3 months before screening and agree to maintain them throughout the study (unless required per the restrictions).
* Agree to follow the restrictions on concomitant treatments.
* Agree to follow the restrictions on lifestyle.
* Agree to avoid pregnancy throughout the study if of childbearing potential by using any preferred contraceptive method.
* Willing and able to agree to the requirements of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

* Individuals who are lactating, planning to become pregnant during the study, or pregnant as confirmed by a positive pregnancy test at Visit 2.
* Have a known sensitivity, intolerability, or allergy to any of the components of the study dietary interventions and/or CGM sensor.
* Have followed a ketogenic, Mediterranean, low-carbohydrate, vegetarian, vegan or any other special diet in the 6 months prior to screening.
* Have been diagnosed with Type I or II diabetes or thyroid disease.
* Have blood pressure of ≥ 160 systolic or ≥ 100 diastolic mmHg.
* Have a history or current diagnosis of eating disorders such as anorexia or bulimia.
* Have current symptoms, or symptoms within the past 7 days, of an acute infection (e.g., fever, respiratory symptoms such as persistent cough or difficulty breathing), that may influence study outcomes as assessed by the investigator.
* Have medical condition(s) known to interfere with absorption, distribution, metabolism, or excretion of protein, fat, or micronutrients (e.g., Crohn's disease, short bowel, acute or chronic pancreatitis, or pancreatic insufficiency).
* Have a history of gallbladder disease (e.g., cholelithiasis, cholecystitis), cholecystectomy, gout, or kidney stones.
* Have a history of heart/cardiovascular disease, renal disease (dialysis or renal failure), hepatic impairment/disease, immune disorders and/or immunocompromised (i.e., HIV/AIDS).
* Have a history of cancer (except localized skin cancer without metastases or in situ cervical cancer) with recovery occurring within 5 years before the screening visit.
* Are receiving treatments for or have been hospitalized in the last 12 months for psychiatric disorders (e.g., depression, bipolar disorder, schizophrenia, etc.).
* Major surgery in 3 months prior to screening or planned major surgery during the study.
* Have a history of alcohol or substance abuse in the 12 months prior to screening (including having been hospitalized for such an in-patient or out-patient intervention program) or use that in the opinion of the investigator may be a concern for the study.
* Current enrollment or past participation in another study with either any product(s) with at least one active ingredient or a dietary intervention, within 28 days before screening or longer, if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study.
* Living in the same household as another currently enrolled participant in the present study.
* Any other medical condition/situation or use of medications/supplements/therapies that, in the opinion of the investigator, may adversely affect the participant's ability to participate in the study or its measures or pose a significant risk to the participant.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-02-03 (Estimated); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of a healthy beef-centric diet on inflammation in a metabolic syndrome (MetS) and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in inflammatory marker composite (combination of hs-CRP, IL-6, IL-10, IL-1β, and TNF-α)

SECONDARY OUTCOMES:
To evaluate the effect of a healthy beef-centric diet on systolic blood pressure (SBP) in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in SBP
To evaluate the effect of a healthy beef-centric diet on diastolic blood pressure (DBP) in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in DBP
To evaluate the effect of a healthy beef-centric diet on body weight in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in body weight
To evaluate the effect of a healthy beef-centric diet on body mass index (BMI) in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in BMI
To evaluate the effect of a healthy beef-centric diet on glucose control (fasting insulin serum) in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in the fasting insulin serum
To evaluate the effect of a healthy beef-centric diet on glucose control (fasting glucose serum) in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in the fasting glucose serum
To evaluate the effect of a healthy beef-centric diet on glycemic patterns in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in mean 72-hour interstitial glucose levels, as assessed by continuous glucose monitoring (CGM) over 3-day periods
To evaluate the effect of a healthy beef-centric diet on quality of life in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in quality of life, as assessed by the Food Benefits Assessment (FBA) Questionnaire on a 5-point Likert Scale: items are scored from 1 (Never / Certainly not) to 5 (Always / Certainly). The scores are transformed on a scale from 0 to 100 with higher scores indicating higher positive impact and/or satisfaction from daily diet.
To evaluate the effect of a healthy beef-centric diet on blood lipids (total cholesterol) in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in the total cholesterol parameter of an advanced lipid profile
To evaluate the effect of a healthy beef-centric diet on blood lipids (high-density lipoprotein (HDL) cholesterol) in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in the HDL cholesterol parameter of an advanced lipid profile
To evaluate the effect of a healthy beef-centric diet on blood lipids (low-density lipoprotein (LDL) cholesterol) in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in the LDL cholesterol parameter of an advanced lipid profile
To evaluate the effect of a healthy beef-centric diet on blood lipids (HDL:LDL ratio) in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in the HDL:LDL ratio parameter of an advanced lipid profile
To evaluate the effect of a healthy beef-centric diet on blood lipids (triglycerides) in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in the triglycerides parameter of an advanced lipid profile
To evaluate the effect of a healthy beef-centric diet on blood lipids (apolipoprotein B (ApoB)) in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in the ApoB parameter of an advanced lipid profile
To evaluate the effect of a healthy beef-centric diet on blood lipids (lipid fraction) in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in the lipid fraction parameter of an advanced lipid profile
To evaluate the effect of a healthy beef-centric diet on short-term average glucose control in a MetS and/or pre-diabetic population, compared to a healthy U.S.-style dietary pattern | Baseline to Week 5
  Change from baseline to Week 5 in average blood glucose, as assessed by fructosamine levels

OTHER OUTCOMES:
To evaluate the effect of a healthy beef-centric diet and a healthy U.S.-style dietary pattern on total caloric intake | Baseline to Week 5
  Change from baseline to Week 5 in total caloric intake
To assess the safety (vital signs) of the healthy beef-centric diet | Baseline to Week 5
  Vital signs (heart rate [HR])
To assess the safety of the healthy beef-centric diet (Hemoglobin) | Baseline to Week 5
  Safety Laboratory Parameters - Hematology Parameters (Hemoglobin)
To assess the safety of the healthy beef-centric diet (Hematocrit) | Baseline to Week 5
  Safety Laboratory Parameters - Hematology Parameters (Hematocrit)
To assess the safety of the healthy beef-centric diet (White Blood Cell (WBC) count) | Baseline to Week 5
  Safety Laboratory Parameters - Hematology Parameters (WBC count with differentials: neutrophils, eosinophils, basophils, lymphocytes, monocytes)
To assess the safety of the healthy beef-centric diet (Red Blood Cell (RBC) count) | Baseline to Week 5
  Safety Laboratory Parameters - Hematology Parameters (RBC Count)
To assess the safety of the healthy beef-centric diet (Red Blood Cell Distribution Width (RCDW)) | Baseline to Week 5
  Safety Laboratory Parameters - Hematology Parameters (RCDW)
To assess the safety of the healthy beef-centric diet (Mean Corpuscular Volume (MCV)) | Baseline to Week 5
  Safety Laboratory Parameters - Hematology Parameters, RBC Index - MCV
To assess the safety of the healthy beef-centric diet (Mean Corpuscular Hemoglobin (MCH)) | Baseline to Week 5
  Safety Laboratory Parameters - Hematology Parameters, RBC Index - MCH
To assess the safety of the healthy beef-centric diet (Mean Corpuscular Hemoglobin Concentration (MCHC)) | Baseline to Week 5
  Safety Laboratory Parameters - Hematology Parameters, RBC Index - MCHC
To assess the safety of the healthy beef-centric diet (Platelet count) | Baseline to Week 5
  Safety Laboratory Parameters - Hematology Parameters (Platelet count)
To assess the safety of the healthy beef-centric diet (Mean Platelet Volume (MPV)) | Baseline to Week 5
  Safety Laboratory Parameters - Hematology Parameters (MPV)
To assess the safety of the healthy beef-centric diet (Blood smear) | Baseline to Week 5
  Safety Laboratory Parameters - Hematology Parameters (Blood smear)
To assess the safety of the healthy beef-centric diet (Sodium) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (Sodium)
To assess the safety of the healthy beef-centric diet (Potassium) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (Potassium)
To assess the safety of the healthy beef-centric diet (Chloride) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (Chloride)
To assess the safety of the healthy beef-centric diet (Blood urea nitrogen (BUN)) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (BUN)
To assess the safety of the healthy beef-centric diet (Creatinine) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (Creatinine)
To assess the safety of the healthy beef-centric diet (Estimated glomerular filtration rate (eGFR)) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (eGFR)
To assess the safety of the healthy beef-centric diet (Total protein) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (Total protein)
. To assess the safety of the healthy beef-centric diet (Albumin) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (Albumin)
To assess the safety of the healthy beef-centric diet (Globulin) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (Globulin)
To assess the safety of the healthy beef-centric diet (Total bilirubin) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (Total bilirubin)
To assess the safety of the healthy beef-centric diet (Fasted glucose) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (Fasted glucose)
To assess the safety of the healthy beef-centric diet (Alanine transaminase (ALT)) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (ALT)
To assess the safety of the healthy beef-centric diet (Aspartate transaminase (AST)) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (AST)
To assess the safety of the healthy beef-centric diet (Alkaline phosphatase (ALP)) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (ALP)
To assess the safety of the healthy beef-centric diet (Gamma glutamyl transferase (GGT)) | Baseline to Week 5
  Safety Laboratory Parameters - Clinical Chemistry Parameters (GGT)
To assess the safety of the healthy beef-centric diet (adverse event reports) | Baseline to Week 5
  Reports of adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Shalene McNeill, Study Chair — National Cattlemen's Beef Association (NCBA), a contractor to the Beef Checkoff
Locations (1):
- Apex Trials, Guelph, Ontario - on, Canada

IPD SHARING:
Plan to Share IPD: No